CLINICAL TRIAL: NCT01577511
Title: Invasiveness and Chemoresistance of Cancer Stem Cells in Colon Cancer: Molecular Characterization and Implications for Therapeutic Strategies
Brief Title: Invasiveness and Chemoresistance of Cancer Stem Cells in Colon Cancer
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/JFB-01; 2011-A01141-40 (Other: ANSM)
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Neoplasms
Keywords: invasive potential; molecular characterisation of circulating cells
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peroperative blood sample plus primary and metastatic tumor biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 30 Patients: Patients with operable, stage III or IV, adenocarcino-type colorectal cancer treated at the Nîmes University Hospital.
  Intervention: Samples and follow up
  Interventions: Biological: Samples and follow up

INTERVENTIONS:
Biological: Samples and follow up — Samples: Peroperative blood sample plus primary and metastatic tumor biopsies.
  Follow-up: disease outcomes assessed at 24 months

SUMMARY:
The main objective of this study is to identify and characterize subpopulations of cells with invasive capacity in colorectal cancer from primary tumor, blood and metastatic samples.

DETAILED DESCRIPTION:
Secondary objectives include:

* Determine the intrinsic properties essential for the dissemination and chemoresistance of these cells capable of initiating tumors
* Identify a "molecular signature" for potential invasiveness and chemoresistance of cells initiating metastases.
* Describe the evolution of patients during 24 months of follow up and correlations with observed cellular profiles.
* Enrich the tumor bank of the institution.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient with adenocarcinoma-type colorectal cancer:
* stage III at diagnosis, surgical resection of the primary tumor proposed.
* stage IV at diagnosis, surgical resection of the primary tumor and possibly of metastases proposed.
* Stage IV who have already undergone surgical excision of the primary tumor, and for whom metastasectomy is now proposed.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patients for whom surgical resection of the primary tumor is not considered as an option
* PStage IV at diagnosis, but metastasectomy is not considered as an option
* Patients with positive HIV, Hepatitis B or Hepatitis C serology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable, stage III or IV, adenocarcino-type colorectal cancer treated at the Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Ability to maintain the cells isolated from colorectal tumors in culture or 3D collagen matrices and then infect these cells to make them express reporter genes: yes/no. | Baseline (Day 0)

SECONDARY OUTCOMES:
Serology HIV | baseline; day 0
Serology Hepatitis B | baseline; day 0
Serology Hepatitis C | baseline; day 0
Location of primary tumor | base line; day 0
  right colon, left colon, transverse colon, sigmoid, rectum
Age at diagnosis | baseline, day 0
Metastases from the outset: Yes / No | baseline, day 0
Resection proposed: yes/no | baseline, day 0
Chemotherapy proposed? yes/no | baseline, day 0
Number of metastases | 24 months
Resection performed: yes/no | 24 months
Number of chemotherapy sessions performed | 24 months
Objective tumoral response to treatment? yes/no | 24 months
Tumor recurrence: yes/no | 24 months
Vital status | 24 months
  living/deceased
Ability to establish tumor xenografts from injected cells: yes/no. | baseline; Day 0
Ability to detect subpopulations of tumor cells expressing fluorophores by flow cytometry after isolation: yes/no | baseline; day 0
Characterization of mRNA expression profiling and micro-RNA + in vitro EMT cells | baseline; day 0
World Health Organisation Score | 24 months
Tumor staging | 24 months
Number of surgeries performed | 24 months
Number of circulating cancer cells per ml blood | baseline; day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Bourgaux, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France

REFERENCES:
- [Result] Grillet F, Bayet E, Villeronce O, Zappia L, Lagerqvist EL, Lunke S, Charafe-Jauffret E, Pham K, Molck C, Rolland N, Bourgaux JF, Prudhomme M, Philippe C, Bravo S, Boyer JC, Canterel-Thouennon L, Taylor GR, Hsu A, Pascussi JM, Hollande F, Pannequin J. Circulating tumour cells from patients with colorectal cancer have cancer stem cell hallmarks in ex vivo culture. Gut. 2017 Oct;66(10):1802-1810. doi: 10.1136/gutjnl-2016-311447. Epub 2016 Jul 25. PMID 27456153